CLINICAL TRIAL: NCT03338959
Title: A Pilot Study of Pembrolizumab and Neoadjuvant Radiation for Large, High-Risk Soft Tissue Sarcomas
Brief Title: Pembrolizumab and Radiation Therapy in Treating Patients With Intermediate or High-Grade Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lee Cranmer, Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9661; NCI-2017-01933 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9661 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9217020 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Soft Tissue Sarcoma; Recurrent Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, radiation therapy) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for 3 months in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy daily for 5-6 weeks.
  Interventions: Biological: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation; NOS; Energy Type

SUMMARY:
This phase I/II trial studies pembrolizumab and radiation therapy in treating patients with intermediate or high-grade soft tissue sarcoma. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving pembrolizumab and radiation therapy may work better in treating patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive pembrolizumab intravenously (IV) per institutional standard at the Seattle Cancer Care Alliance as an outpatient therapy. Cycles repeat every 3 weeks, up to a maximum of three doses, for 3 months in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy daily for 5-6 weeks beginning on Day 1 of Week 2.

After completion of study treatment, patients are followed up at 30 days after last dose, 90 days after last dose, 30 days after post-operative visit (wound care follow-up), and then every 12 weeks for up to 1 year, then every 6 months up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Be ≥18 years of age on day of signing informed consent documents
* Have measurable disease based on RECIST 1.1
* Have newly diagnosed disease or localized recurrent or oligometastatic lesions that are candidates for radiation

  * NOTE: Subjects may not have any prior systemic therapy or radiation for this sarcoma. They may have received systemic therapy and/or radiation for a different cancer
  * NOTE: Oligometastatic disease will be defined as 3 or fewer detectable lesions with plans to radiate all detectable disease with conventionally fractionated radiation prior to resection
* Have an intermediate- or high-grade soft tissue sarcoma at the discretion of the reviewing Sarcoma pathologist
* The tumor must be at least 3 cm in maximum dimension for intermediate-grade tumors, or 1.5 cm in maximum dimension for high-grade tumors
* Have plans to undergo neo-adjuvant radiation and surgery with curative intent. A minimum of 45 Gy is necessary, planned to be administered over a minimum of 25 fractions
* Be willing to provide tissue from a newly obtained core incisional or excisional biopsy of a tumor lesion. Archival tissue from a recent clinical or research biopsy (within 90 days prior to Week 1 treatment) may be used in place of a fresh tissue biopsy
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale or > 70% on the Karnofsky scale. Evaluation of performance status is to be performed within 7 days prior to the date of enrollment
* Absolute neutrophil count (ANC) >= 1,500/mcL (performed within 28 days of enrollment)
* Platelets >= 100,000/mcL (performed within 28 days of enrollment)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (performed within 28 days of enrollment)

  * Criteria must be met without erythropoeiten dependency and without packed red blood cell (pRBC) transfusion within last two weeks
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (performed within 28 days of enrollment)

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 28 days of enrollment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN (performed within 28 days of enrollment)
* Albumin >= 2.5 mg/dL (performed within 28 days of enrollment)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 28 days of enrollment)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 28 days of enrollment)
* Female subjects of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication
* All individuals of child-bearing potential must be willing to use an adequate method of contraception, from the first dose of the study medication through 120 days after the last dose of study medication

Exclusion Criteria:

* Has had prior radiation to affected area
* Has one of the following sarcoma subtypes where neoadjuvant chemotherapy is established as practice at our institution: extra-skeletal Ewing's sarcoma, embryonal rhabdomyosarcoma, alveolar rhabdomyosarcoma

  * NOTE: Pleomorphic rhabdomyosarcoma is allowed. Bone sarcomas including osteosarcoma, Ewing's sarcoma and chondrosarcoma are not allowed. Extra-skeletal Osteosarcoma is considered a soft tissue sarcoma and is allowed.
* Has a diagnosis of immunodeficiency or has an active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid)
* Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years

  * NOTE: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
* Has current or a history of any distant metastatic disease (including brain)

  *NOTE: An isolated or oligo-metastatic regional recurrence may be allowed if all other criteria are met, curative attempt is being pursued
* Has known history of (non-infectious) pneumonitis that required steroids, or has current evidence of pneumonitis
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with adherence to the requirements of the trial
* Is pregnant (positive urine pregnancy test within 72 hours prior to enrollment) or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. If a urine pregnancy test is positive or cannot be confirmed negative, a serum pregnancy test will be required
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-CTLA4 or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory 1-cell receptor (eg, CTLA-4, OX 40, CD137)
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) infection
* Has received a live vaccine or live-attenuated vaccine within 30 days of planned start of study therapy. Administration of killed vaccines is allowed. Note: Any licensed coronavirus (COVID-19) vaccine (including for emergency use) is allowed in the study as long as they are messenger ribonucleic acid (mRNA) vaccines, adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy. Investigational vaccines (i.e., those not licensed or approved for emergency use) are not allowed.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate, in the opinion of the treating investigator or has not adequately recovered from any major surgery or has ongoing surgical complications
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
Started | 27
Completed | 9
Not Completed | 18
Not completed — Patients remain in Long-Term Follow-Up | 17
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  Aged Under 18 at Enrollment | 0
  Aged 18-29 at Enrollment | 1
  Aged 30-39 at Enrollment | 1
  Aged 40-49 at Enrollment | 2
  Aged 50-59 at Enrollment | 4
  Aged 60-69 at Enrollment | 9
  Aged 70 and Above at Enrollment | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Tumor Necrosis
Description: Necrosis greater than or equal to 90% at pathologic assessment at time of surgery
Time Frame: From baseline through wound care follow-up visit (up to 8 months)
Population: 24 out of 27 participants evaluable for the primary endpoint. 4 participants experienced necrosis greater than 90%.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
Number analyzed (Participants) | 24
Participants | 4

2. Secondary Outcome: Incidence of Adverse Events
Description: Treatment-related adverse events (AEs) experienced by participants evaluated by Common Terminology Criteria for Adverse Events (CTCAE) 5.0 and determined to be possibly related, probably related, or definitely related to either pembrolizumab therapy, radiation therapy, or both.
Time Frame: Through the wound care follow-up visit (up to 8 months)
Population: All participants evaluable for adverse events.
Measure: Number; unit: events experienced
Groups:
- Grade 1 Events: Treatment-related Grade 1 Adverse Events (AEs) experienced by participants as defined by CTCAE 5.0 criteria.
- Grade 2 Events: Treatment-related Grade 2 Adverse Events (AEs) experienced by participants as defined by CTCAE 5.0 criteria.
- Grade 3 Events: Treatment-related Grade 3 Adverse Events (AEs) experienced by participants as defined by CTCAE 5.0 criteria.
- Grade 4 Events: Treatment-related Grade 4 Adverse Events (AEs) experienced by participants as defined by CTCAE 5.0 criteria.
- Grade 5 Events: Treatment-related Grade 5 Adverse Events (AEs) experienced by participants as defined by CTCAE 5.0 criteria.
Arm/Group | Grade 1 Events | Grade 2 Events | Grade 3 Events | Grade 4 Events | Grade 5 Events
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
events experienced
  Dermatitis Radiation | 12 | 7 | 0 | 0 | 0
  Fatigue | 11 | 3 | 0 | 0 | 0
  Rash maculo-papular | 5 | 3 | 0 | 0 | 0
  Diarrhea | 5 | 1 | 0 | 0 | 0
  Tumor pain | 2 | 2 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 3 | 1 | 0 | 0
  Wound dehiscence | 2 | 1 | 1 | 0 | 0
  Hypothyroidism | 0 | 4 | 0 | 0 | 0
  Nausea | 1 | 2 | 0 | 0 | 0
  Pain in extremity | 1 | 1 | 0 | 0 | 0
  Anorexia | 1 | 1 | 0 | 0 | 0
  Edema limbs | 2 | 0 | 0 | 0 | 0
  Anemia | 0 | 1 | 1 | 0 | 0
  Bullous dermatitis | 2 | 0 | 0 | 0 | 0
  Skin and subcutaneous disorders - Other - Erythema | 2 | 0 | 0 | 0 | 0
  Dizziness | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 1 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 1 | 0 | 0
  Pneumothorax | 1 | 0 | 0 | 0 | 0
  Dry skin | 1 | 0 | 0 | 0 | 0
  Pruritus | 0 | 1 | 0 | 0 | 0
  Dehydration | 0 | 1 | 0 | 0 | 0
  Weight loss | 1 | 0 | 0 | 0 | 0
  Peripheral sensory neuropathy | 1 | 0 | 0 | 0 | 0
  Cough | 1 | 0 | 0 | 0 | 0
  Hypokalemia | 1 | 0 | 0 | 0 | 0
  Peripheral ischemia | 0 | 0 | 0 | 1 | 0
  Chest wall pain | 0 | 1 | 0 | 0 | 0
  Blood and lymphatic system disorders - Other - Eosinophil count increased | 1 | 0 | 0 | 0 | 0
  Thyroid Stimulating Hormone Increased | 1 | 0 | 0 | 0 | 0
  Rectal pain | 1 | 0 | 0 | 0 | 0
  Wound infection | 0 | 0 | 1 | 0 | 0
  Localized edema | 1 | 0 | 0 | 0 | 0
  Urinary urgency | 1 | 0 | 0 | 0 | 0
  Pelvic pain | 1 | 0 | 0 | 0 | 0
  Urinary retention | 0 | 1 | 0 | 0 | 0
  Neuralgia | 1 | 0 | 0 | 0 | 0
  Thromboembolic event | 0 | 1 | 0 | 0 | 0
  Hypomagnesemia | 1 | 0 | 0 | 0 | 0
  Vaginal hemorrhage | 0 | 0 | 1 | 0 | 0
  Colitis | 0 | 1 | 0 | 0 | 0
  Skin and subcutaneous disorders - Other - Rash | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Partial Response Rate
Description: Proportion of patients who achieved a partial response based on modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR.
Time Frame: From baseline through wound care follow-up visit (up to 8 months)
Population: 26 out of 27 participants evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
Number analyzed (Participants) | 26
proportion of participants | 0.08 [0.01 to 0.25]

4. Secondary Outcome: Complete Response Rate
Description: Rate of disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm as defined per RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR.
Time Frame: From baseline through wound care follow-up visit (up to 8 months)
Population: 26 out of 27 participants evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
Number analyzed (Participants) | 26
proportion of participants | 0.00 [0.00 to 0.13]

5. Secondary Outcome: Overall Response Rate
Description: Rate of participants who experienced a Complete Response (CR) + Partial Reponse (PR) as defined per RECIST v1.1 criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR.
Time Frame: From baseline through wound care follow-up visit (up to 8 months)
Population: 26 out of 27 participants evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
Number analyzed (Participants) | 26
proportion of participants | 0.08 [0.01 to 0.25]

ADVERSE EVENTS:
Time Frame: All adverse events will be recorded from the day informed consent is signed through the Wound Care Follow-Up visit (e.g. up to 8 months)
Description: Subjects with an Adverse Event (AE) of Grade >1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anti-neoplastic therapy, whichever occurs first. Serious Adverse Events (SAEs) that occur within 90 days of the last dose of pembrolizumab or 30 days following cessation of pembrolizumab if the participant initiates a new anticancer therapy - whichever is earlier should also be followed and recorded.
Arm/Group | Treatment (Pembrolizumab, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 5/27
Other Adverse Events (participants affected / at risk) | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Radiation Therapy) (N=27)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Acute Transverse Colon Diverticulitis
Hallucinations (Psychiatric disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Radiation Therapy) (N=27)
Fatigue (General disorders) | 17 (18)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 14 (16)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 9 (9)
Anorexia (Gastrointestinal disorders) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (9)
Constipation (Gastrointestinal disorders) | 5 (5)
Presyncope (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5)
Hypothyroidism (Endocrine disorders) | 4 (4)
Lymphocyte count decreased (Investigations) | 3 (7)
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Edema Limbs (General disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Neuralgia (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Bullous dermtitis (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) — Erythema
Pain (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Blurred vision (Eye disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Blister
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Lesion
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Rash
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Scalp lesion
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Skin lesion
Fever (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Phantom pain (Nervous system disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Tendinitis
Sinus bradycardia (Cardiac disorders) | 1 (1)
Investigations - Other (Investigations) | 1 (1) — Eosinophil count increased
Gum infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03338959/Prot_SAP_000.pdf